CLINICAL TRIAL: NCT02059746
Title: Perineal Consequences of Twin Pregnancies According to Mode of Delivery
Acronym: JUMODA-CP
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: AOI/2013/RdeT
Record Dates: First submitted 2014-02-07; First posted 2014-02-11 (Estimated); Last update posted 2025-11-19 (Actual); Status verified 2016-04

CONDITIONS: Pregnancy, Multiple
Keywords: cesarean section; vaginal birth; twins; urinary incontinence; sexuality; quality of life
MeSH Terms: conditions — Urinary Incontinence; Sexuality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Vaginal birth: Patients in the group give birth vaginally.
  Intervention: Questionnaires sent by mail
  Interventions: Other: Questionnaires sent by mail
- Cesaren section: Patients in this group give birth via cesarean section.
  Intervention: Questionnaires sent by mail
  Interventions: Other: Questionnaires sent by mail

INTERVENTIONS:
Other: Questionnaires sent by mail — The questionnaires necessary for the study are mailed to patients at 3 and 12 months post-partum.

SUMMARY:
This is an ancillary study to the "JUMODA" (National Prospective and Comparative Study on the Mode of Delivery of Twins) study: please see NCT01987063.

The main objective of this study is to investigate the role of the mode of delivery (vaginal versus cesarean) as a risk factor for the occurrence of urinary incontinence at 3 months post-delivery in primiparous women delivering twins after 34 weeks of pregnancy.

DETAILED DESCRIPTION:
The secondary objectives of this study are to compare the following elements between primiparous mothers giving birth to twins vaginally versus by caesarean section after 34 weeks of pregnancy (comparisons will be made at 3 months ant at 12 months post-partum):

A. Diagnosis, type and severity of urinary incontinence via the ICIQ-UI questionnaire

B. Urinary, anorectal and perineal symptoms via the PFDI-20 questionnaire

C. Quality of life related to urinary, anorectal and pelvic floor symptoms via the PFIQ-7 questionnaire

D. Sexuality via the PISQ-12 questionnaire

E. General quality of life via the SF-12 questionnaire

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient is available for 12 months of follow-up following delivery
* The patient was included in the JUMODA study
* Primiparous
* Birth of 2 live children after 34 weeks of pregnancy

Exclusion Criteria:

* Adult patient under guardianship
* Patient under judicial protection
* It proves impossible to correctly inform the patient
* Birth occurring before 34 weeks of pregnancy
* Birth not resulting in 2 living children

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is an ancillary to the "JUMODA" study (please see NCT01987063). The study population is composed of primiparous women pregnant with twins (non primiparous patients in the study JUMODA will therefore not includable), giving birth after 34 weeks to 2 live children.
Sampling Method: Non-Probability Sample
Enrollment: 3039 (Actual)
Dates: Start 2014-02; Primary Completion 2015-03-01 (Actual); Study Completion 2016-03-01 (Actual)

PRIMARY OUTCOMES:
Presence/absence of urinary incontinence | 3 months post-partum
  Defined by a response of 1 to 5 on the first question of the ICIQ-UI questionnaire.

SECONDARY OUTCOMES:
The ICIQ-UI questionnaire | 3 months post-partum
  ICIQ-Urinary Incontinence Form
The PFDI-20 questionnaire | 3 months post-partum
The ICIQ-UI questionnaire | 12 months post-partum
  ICIQ-Urinary Incontinence Form
The PFDI-20 questionnaire | 12 months post-partum
The PFIQ-7 questionnaire | 3 months post-partum
The PFIQ-7 questionnaire | 12 months post-partum
The PISQ-12 questionnaire | 3 months post-partum
The PISQ-12 questionnaire | 12 months post-partum
The SF-12 questionnaire | 3 months post-partum
The SF-12 questionnaire | 12 months post-partum

CONTACTS AND LOCATIONS:
Overall Officials: Renaud de Tayrac, MD, PhD, Study Director — Centre Hospitalier Universitaire de Nîmes
Locations (2):
- France (2):
  - CHRU de Montpellier - Hôpital Arnaud de Villeneuve, Montpellier
  - CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes

REFERENCES:
- [Result] Bechard F, Castelli C, Alonso S, Vintejoux E, Goffinet F, Letouzey V, Schmitz T, de Tayrac R. Impact of mode of delivery of twins on the pelvic floor 3 and 12 months post-partum-part II. Int Urogynecol J. 2019 Jun;30(6):893-899. doi: 10.1007/s00192-018-3785-1. Epub 2018 Oct 5. PMID 30291380